CLINICAL TRIAL: NCT00670254
Title: Placebo-controlled, Randomised, Double-blind Study to Investigate the Efficacy and Safety of Low Dose Hydrocortisone to Prevent the Development of Septic Shock in Patients With Severe Sepsis
Brief Title: Hydrocortisone for Prevention of Septic Shock
Acronym: HYPRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); SepNet - Critical Care Trials Group (Other); Coordination Centre for Clinical Trials Leipzig (Unknown)
Responsible Party: Principal Investigator, Didier Keh, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYPRESS; 01KG0701 (Other: BMBF); 2007-004401-10 (EudraCT Number)
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Severe Sepsis
Keywords: Sepsis; Septic; Shock; Glucocorticoids; Hydrocortisone
MeSH Terms: conditions — Sepsis; Shock | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone (Experimental)
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Application is identical to experimental arm
  Arms: Placebo
Drug: Hydrocortisone — 50 mg loading dose, continuous infusion of 200 mg/d for 5 d, 100 mg/d for 2d, 50 mg/d for 2 d, and 25 mg/d for 2 d.
  Arms: Hydrocortisone

SUMMARY:
Severe sepsis is a disease with a high mortality. Development of shock is a most serious complication and increases the risk of death considerably. Application of low dose hydrocortisone is currently recommended only in patients after severe septic shock has been established. Hydrocortisone therapy has a hemodynamic stabilizing effect and may reverse shock, however, the preventive application has not been investigated in a larger study. The study investigates whether low dose hydrocortisone prevents the development of shock in patients with severe sepsis. It is postulated that shock prevention may also affect morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Severe sepsis according to ACCP/CCM criteria
* Onset of severe sepsis < 48 hours
* Informed consent
* Effective contraception in fertile women

Exclusion Criteria:

* Septic shock
* Known hypersensitivity to hydrocortisone and additives
* Glucocorticoid history which warrants continuation of glucocorticoid administration
* Other indication for systemic glucocorticoid therapy
* DNR-order
* Moribund patient
* Pregnancy
* Breast feeding women
* Age < 18 years
* Other interventional study
* Relationship to investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2009-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Septic shock | 14 days

SECONDARY OUTCOMES:
Mortality | 28, 90, and 180 days; ICU and hospital
Length of stay | ICU and hospital (3-6 months)
Time to death | 28, 90, and 180 days
Time to septic shock | 14 days
Mechanical ventilation | until ICU discharge
Renal replacement therapy | until ICU discharge
Organ dysfunction (SOFA score) | until ICU discharge but day 14 at maximum
Frequency of weaning failure | until ICU discharge
Frequency and severity of muscle weakness | until ICU discharge
Frequency of gastrointestinal bleeding | 28 days
Frequency of secondary infections | 28 days
Delir | ICU discharge
Hypernatremia | 14 days
Hyperglycemia | 14 days
Other adverse events | 28 days
Posttraumatic stress disorder / health-related quality of life | Hosptal discharge and 180 days after hospital discharge
Immune response to hydrocortisone | 6 days
Adrenal function | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Reinhart, MD, Principal Investigator — University Hospital Jena; Dept. of Anesthesiology an Intensive Care Medicine; Didier Keh, MD, Study Chair — Charité Universitaetsmedizin Berlin, Dept. of Anesthsiology and Intensive Care Medicine; Frank M Brunkhorst, MD, Study Director — University Hospital Jena, Dept. of Anesthesiology and Intensive Care Medicine; Markus Loeffler, MD, Study Director — University Leipzig, Coordination Center of Clinical Studies (KKSL)
Locations (30):
- Germany (30):
  - Universitaetsklinikum Aachen, Operative Intensivmedizin Erwachsene, Aachen
  - Zentralklinik Bad Berka GmbH, Zentrum für Anaesthesie, Intensivtherapie und Notfallmedizin, Bad Berka
  - HELIOS Klinikum Bad Saarow; Zentrum für Anaesthesiologie, Intensivmedizin, Notfallmedizin und Schmerztherapie, Bad Saarow
  - St. Joseph Krankenhaus, Institut fue Anaesthesie, Schwerpunkt operative Intensivmedizin und SchmerztherapieAnaesthesie, operative Intensiv- und Notfallmedizin, Berlin
  - Vivantes Auguste-Viktoria-Klinikum, Klinik fuer Anaesthesiologie, Intensivmedizin und Schmerztherapie, Berlin
  - Vivantes Klinikum Neukoelln,Klinik fuer Innere Medizin, Kardiologie und konservative Intensivmedizin, Berlin
  - Vivantes Klinikum-Neukoelln, Klinik fuer Anaesthesie, operative Intensivmedizin und Schmerztherapie, Berlin
  - Vivantes Klinikum Hellersdorf, Klinik fuer Anaesthesie, operative Intensivmedizin und Schmerztherapie, Berlin
  - Helios Klinikum Berlin Buch, Klinik für Intensivmedizin, Berlin
  - Charité Universitaetsmedizin Berlin, Campus Virchow-Klinikum und Campus Mitte, Med. Klinik mit Schwerpunkt Infektiologie und Pneumologie, Berlin
  - Charité Universitaetsmedizin Berlin, Campus Virchow-Klinikum und Mitte Klinik für Anaesthesiologie und operative Intensivmedizin, Berlin
  - Charité Universitätsmedizin Berlin, Campus Virchow-Klinikum, Med. Klinik mit Schwerpunkt Nephrologie und internistische Intensivmedizin, Berlin
  - Vivantes Humboldt-Klinikum, Klinik für Innere Medizin - Kardiologie und konservative Intensivmedizin, Berlin
  - Rheinische Friedrich-Wilhelms-Universitaet, Klinik für Anaesthesiologie und Operative Intensivmedizin, Bonn
  - St. Elisabeth-Krankenhaus Köln-Hohenlind, Klinik für Anaesthesiologie und operative Intensivmedizin, Cologne
  - Kliniken der Stadt Koeln - Krankenhaus Merheim, Klinik für Anaesthesiologie und operative Intensivmedizin, Cologne
  - Krankenhaus Dresden-Friedrichstadt, Klinik für Anaesthesiologie und Intensivmedizin, Dresden
  - Universitaetsklinik Carl Gustav Carus Dresden, Dresden
  - Helios Klinikum Erfurt, Klinik fuer Anaesthesie, Intensivmedizin und Schmerztherapie, Erfurt
  - Universitaetsklinikum Freiburg, Anaesthesiologische Universitaetsklinik - Abteilung Anaesthesiologie und Intensivtherapie, Freiburg im Breisgau
  - Ernst Moritz Arndt Universitaet Greifswald, Klinik und Poliklinik für Anaesthesiologie und Intensivmedizin, Greifswald
  - Medizinische Fakultaet der Martin-Luther-Universitaet Halle-Wittenberg - Universitaetsklinikum Halle (Saale), Halle
  - Krankenhaus Martha-Maria Halle-Doelau GmbH, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Klinik für Intensivmedizin, Hamburg
  - Klinikum Heidenheim, Klinik für Anaesthesiologie und operative Intensivmedizin, Heidenheim
  - Klinik Henningsdorf der Oberhavel-Kliniken GmbH, Abteilung für Anaesthesie und Intensivmedizin, Henningsdorf
  - Friedrich Schiller Universität, Klinik für Anaesthesiologie und Intensivmedizin, Jena
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Klinik für Anaesthesiologie und Operative Intensivmedizin, Kiel
  - Universitaetsklinikum Leipzig AöR, Klinik und Poliklinik für Anaesthesiologie und Intensivtherapie, Leipzig
  - Klinikum Oldenburg GmbH, Klinik fuer Anaesthesiologie, Intensivmedizin, Notfallmedizin und Schmerztherapie, Oldenburg

REFERENCES:
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Reinhart K, Brunkhorst F, Bone H, Gerlach H, Grundling M, Kreymann G, Kujath P, Marggraf G, Mayer K, Meier-Hellmann A, Peckelsen C, Putensen C, Quintel M, Ragaller M, Rossaint R, Stuber F, Weiler N, Welte T, Werdan K; Deutschen Interdisziplinaren Vereinigung fur Intensiv- und Notfallmedizin (DIVI); Deutschen Sepsis-Gesellschaft e.V. (DSG). [Diagnosis and therapy of sepsis. Guidelines of the German Sepsis Society Inc. and the German Interdisciplinary Society for Intensive and Emergency Medicine]. Internist (Berl). 2006 Apr;47(4):356, 358-60, 362-8, passim. doi: 10.1007/s00108-006-1595-x. German. PMID 16532281
- [Background] Engel C, Brunkhorst FM, Bone HG, Brunkhorst R, Gerlach H, Grond S, Gruendling M, Huhle G, Jaschinski U, John S, Mayer K, Oppert M, Olthoff D, Quintel M, Ragaller M, Rossaint R, Stuber F, Weiler N, Welte T, Bogatsch H, Hartog C, Loeffler M, Reinhart K. Epidemiology of sepsis in Germany: results from a national prospective multicenter study. Intensive Care Med. 2007 Apr;33(4):606-18. doi: 10.1007/s00134-006-0517-7. Epub 2007 Feb 24. PMID 17323051
- [Background] Sprung CL, Annane D, Keh D, Moreno R, Singer M, Freivogel K, Weiss YG, Benbenishty J, Kalenka A, Forst H, Laterre PF, Reinhart K, Cuthbertson BH, Payen D, Briegel J; CORTICUS Study Group. Hydrocortisone therapy for patients with septic shock. N Engl J Med. 2008 Jan 10;358(2):111-24. doi: 10.1056/NEJMoa071366. PMID 18184957
- [Background] Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y. Corticosteroids for treating severe sepsis and septic shock. Cochrane Database Syst Rev. 2004;(1):CD002243. doi: 10.1002/14651858.CD002243.pub2. PMID 14973984
- [Background] Keh D, Boehnke T, Weber-Cartens S, Schulz C, Ahlers O, Bercker S, Volk HD, Doecke WD, Falke KJ, Gerlach H. Immunologic and hemodynamic effects of "low-dose" hydrocortisone in septic shock: a double-blind, randomized, placebo-controlled, crossover study. Am J Respir Crit Care Med. 2003 Feb 15;167(4):512-20. doi: 10.1164/rccm.200205-446OC. Epub 2002 Nov 8. PMID 12426230
- [Background] American College of Chest Physicians/Society of Critical Care Medicine Consensus Conference: definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. Crit Care Med. 1992 Jun;20(6):864-74. PMID 1597042
- [Derived] Briegel J, Mohnle P, Keh D, Lindner JM, Vetter AC, Bogatsch H, Lange D, Frank S, Hinske LC, Annane D, Vogeser M; SepNet Critical Care Trials Group. Corticotropin-stimulated steroid profiles to predict shock development and mortality in sepsis: From the HYPRESS study. Crit Care. 2022 Nov 7;26(1):343. doi: 10.1186/s13054-022-04224-5. PMID 36345013
- [Derived] Keh D, Trips E, Marx G, Wirtz SP, Abduljawwad E, Bercker S, Bogatsch H, Briegel J, Engel C, Gerlach H, Goldmann A, Kuhn SO, Huter L, Meier-Hellmann A, Nierhaus A, Kluge S, Lehmke J, Loeffler M, Oppert M, Resener K, Schadler D, Schuerholz T, Simon P, Weiler N, Weyland A, Reinhart K, Brunkhorst FM; SepNet-Critical Care Trials Group. Effect of Hydrocortisone on Development of Shock Among Patients With Severe Sepsis: The HYPRESS Randomized Clinical Trial. JAMA. 2016 Nov 1;316(17):1775-1785. doi: 10.1001/jama.2016.14799. PMID 27695824
- See also: Competence Network Sepsis (SepNet) — http://www.sepsis-gesellschaft.de/DSG/Englisch/SepNet?sid=oKhUu07XmwBjbeKacHsxr0&iid=2